CLINICAL TRIAL: NCT02300545
Title: A Phase II Study of Pazopanib as Front-Line Therapy in Patients With Non-Resectable or Metastatic Soft Tissue Sarcomas Who Are Not Candidates for Chemotherapy
Brief Title: Pazopanib as Front-Line Therapy in Patients With Non-Resectable or Metastatic Soft Tissue Sarcomas Who Are Not Candidates for Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201501057
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Sarcoma, Soft Tissue; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pazopanib (Experimental): Pazopanib will be started at a dose of 200 mg BID for four days, then escalated to a dose of 400 mg BID for four days, then escalated once more to a dose of 800 mg QD for the duration of participation (or until dose reduction, if necessary). Pazopanib should be taken orally without food at least one hour before or two hours after a meal. One cycle of pazopanib is 28 days.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib
  Other Names: GW786034; Votrien

SUMMARY:
Pazopanib is FDA approved as a second line and beyond treatment for metastatic soft tissue sarcoma. There is a population of elderly and debilitated soft tissue sarcoma patients that are not fit for standard first line chemotherapy that is doxorubicin based. As pazopanib is well tolerated with minimal side effects, the investigators propose a phase II study to evaluate pazopanib as a first-line agent in patients with non-resectable or metastatic disease who are not candidates for cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of nonresectable or metastatic soft tissue sarcoma. The following histologies are excluded: embryonal rhabdomyosarcoma, chondrosarcoma, osteosarcoma, Ewing tumors, primitive neuroectodermal tumors, gastrointestinal stromal tumors, dermatofibrosarcoma protuberans, inflammatory myofibroblastic sarcoma, and mixed mesodermal tumors of the uterus.
* Evaluable disease by imaging or physical exam OR measurable disease defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Not a candidate for chemotherapy as determined by treatment physician
* Age ≥ 18 years
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * PT or INR ≤ 1.2 x IULN (if not receiving anticoagulation therapy)
  * PTT ≤ 1.2 x IULN (if not receiving anticoagulation therapy)
  * Total bilirubin ≤ 1.5 x IULN or ≤ 3.0 x IULN with normal AST and ALT in patients with Gilbert's disease
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 30 mL/min/1.73 m2 for patients with creatinine levels above 1.5 mg/dL
  * UPC < 1 or, if UPC ≥ 1, 24-hour urine protein < 1 g; use of urine dipstick for renal function assessment is not acceptable.

Notes:

Subjects may not have had a transfusion within 7 days of screening assessments. Concomitant elevation of bilirubin and AST/ALT above the IULN is not allowed.

Patients receiving anticoagulation therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.

* Ability to swallow and retain oral tablets.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Eligible for cytotoxic chemotherapy.
* Prior systemic therapy for this type of sarcoma. Neoadjuvant or adjuvant therapy more than two years prior would not apply.
* Prior treatment with any VEGFR tyrosine kinase inhibitor.
* Administration of any non-oncologic investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the first dose of pazopanib.
* Use of a strong CYP3A4 inhibitor less than 14 days prior to initiation of study treatment
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Known brain metastases.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib or other agents used in the study.
* Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity (except alopecia).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled seizure disorder, or psychiatric illness/social situations that would limit compliance with study requirements.
* Corrected QT interval (QTc) > 480 msecs.
* History of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina pectoris, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure as defined by the New York Heart Association
* Poorly controlled hypertension (defined as systolic blood pressure of ≥ 140 mmHg or diastolic blood pressure of ≥ 90 mmHg). Note: initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure must be reassessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between antihypertensive medication initiation or adjustment and blood pressure measurement. These three values should be averaged to obtain the mean diastolic and systolic blood pressures, which must be < 140/90 mmHg in order for a patient to be eligible for the study.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding, including (but not limited to) active peptic ulcer disease, known intraluminal metastatic lesions with risk of bleeding, inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other GI conditions with increased risk of perforation, history of abdominal fistula or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Clinically significant gastrointestinal abnormalities that may affect absorption of pazopanib, including (but not limited to) malabsorption syndrome or major resection of the stomach or small bowel.
* History of cerebrovascular accident including transient ischemic attack, pulmonary embolism (PE) (including asymptomatic or previously treated PE), or untreated deep venous thrombosis within the past 6 months. Patients with DVT who are being treated with therapeutic anti-coagulating agents are eligible.
* Major surgery or trauma within 28 days prior to first dose of pazopanib and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage. Note: lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions). Large protruding endobronchial lesions in the mail or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed. Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of thee bronchi are allowed.
* Recent hemoptysis (≥ ½ teaspoon of red blood within 8 weeks before first dose of pazopanib).
* Pregnant and/or breastfeeding. Patient must have a negative serum pregnancy test within 14 days of study entry.
* Known HIV-positivity. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Van Tine, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (7):
- United States (7):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 04/08/2015 and closed to participant enrollment on 02/20/2019.
Period: Overall Study
Arm/Group | Pazopanib
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 78.7 [60 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 40
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate = complete response (CR) + partial response (PR) + stable disease (SD)
  * CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 56
Participants | 22

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Until disease progression (median follow-up of 10.83 months with full range 0.787-42.26 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 56
months | 3.67 [2.62 to 7.25]

3. Secondary Outcome: Overall Survival (OS)
Time Frame: Until death (median follow-up of 10.83 months with full range 0.787-42.26 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 56
months | 14.16 [8.46 to NA] — The upper 95% confidence interval was not reached.

4. Secondary Outcome: Median Overall Change in Quality of Life
Description: * Quality of life will be measured using the Functional Assessment of Cancer Therapy-General (FACT-G7) validated survey
  * 7 statements where the participant can indicate 0 (not at all) up to 4 (very much). The statements include 1) I have lack of energy; 2) I have pain; 3) I have nausea; 4) I worry that my condition will get worse; 5) I am sleeping well; 6) I am able to enjoy life; 7) I am content with the quality of my life right now.
  * The first 4 statements will negatively affect the total score and the last 3 statements will positively affect the total score
  * Each item is scored and then added together, multiplied by 7, and divided by the number of items
  * Total score calculation ranges from 0-28. The higher the score, the better the quality of life
Time Frame: Change from baseline to end of treatment (median length of treatment 70 days (5-515 days)))
Measure: Median (95% Confidence Interval); unit: points on a scale
Arm/Group | Pazopanib
Number analyzed (Participants) | 56
points on a scale | 2 [0.7356979 to 4.5834510]

5. Secondary Outcome: Clinical Outcome Associated With Serum sVEGFR2 Levels (Serum Levels of sVEGFR2 at Each Time Point Will Plotted and Pearson or Spearman's Correlation Coefficient)
Description: The serum levels of sVEGFR2 at each time point will plotted and Pearson or Spearman's correlation coefficient will be calculated to explore their relationship.
Time Frame: From baseline through completion of treatment
Population: There was no funding to process the serum levels of sVEGFR2.
Arm/Group | Pazopanib
Number analyzed (Participants) | 0

6. Secondary Outcome: Clinical Outcome Associated With Serum PICG Levels (Serum Levels of PIGF at Each Time Point Will Plotted and Pearson or Spearman's Correlation Coefficient)
Description: The serum levels of PIGF at each time point will plotted and Pearson or Spearman's correlation coefficient will be calculated to explore their relationship.
Time Frame: From baseline through completion of treatment
Population: There was no funding to process the serum levels of PIGF.
Arm/Group | Pazopanib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: -Reportable adverse events were tracked for 30 days following the last day of study treatment. Median treatment length was 70 days (5 days-515 days). As of first reporting of results, one participant is still receiving treatment.
Description: The adverse events listed in the other (not including serious) adverse event module are deemed to be related to treatment.
Arm/Group | Pazopanib
All-Cause Mortality (participants affected / at risk) | 24/56
Serious Adverse Events (participants affected / at risk) | 27/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=56)
Acute coronary syndrome (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Bowel infarction related to disease (Gastrointestinal disorders) | 1
Colonic fistula (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
GI bleed (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Bronchial infection (Infections and infestations) | 1
Colitis (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 1
Intratumoral hemorrhage (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=56)
Anemia (Blood and lymphatic system disorders) | 18
Chest pain - cardiac (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Blurred vision (Eye disorders) | 3
Vision changes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 10
Belching (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 29
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 27
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 19
Chills (General disorders) | 1
Edema face (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 33
Hair depigmentation (General disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 13
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 21
Blood bilirubin increased (Investigations) | 11
Creatinine increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
GGT increased (Investigations) | 2
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 17
Weight loss (Investigations) | 8
White blood cell decreased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 13
Headache (Nervous system disorders) | 8
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Right hand paralysis (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Night sweats (Reproductive system and breast disorders) | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 23
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT02300545/Prot_SAP_000.pdf